



## NEUROLOGISCHE KLINIK UND POLIKLINIK MIT FRIEDRICH-BAUR-INSTITUT



Direktorin: Prof. Dr. med. M. Dieterich

in Assoziation mit dem Institut für Neuroimmunologie und dem Institut für Schlaganfall- und Demenzforschung

Klinikum der Universität München – Großhadern Neurologische Klinik, Marchioninistr. 15 · D-81377 München

Herrn Prof. Dr. W. Eisenmenger Chairman of the Ethics committee at the Ludwigs-Maximilians-University Pettenkoferstr. 8 80336 München Dr. med. M. Empl

Telefon +49 (0)89 7095 - 3690 Telefax +49 (0)89 7095 - 3677 Neurologische Poliklinik

www.neurologie.klinikum.unimuenchen.de

Postanschrift: Marchioninistr. 15 D-81377 München

Ihr Zeichen: Unser Zeichen: München, den 22.10.2015

Dr. M. Empl

Application to the Ethics Committee for a non-AMG/non-MPG study
Introvision in migraines and headaches - IntroMig

Dear Prof. Eisenmenger,

I have been working for many years in the Headache Department and in the headache outpatient clinic with Prof. Straube and I am planning a study on Introvision in migraines and headache patients. Introvision is a mental self-regulation method which uses a mindfulness technique that was developed by Frau Prof. Wagner, University of Hamburg. It not only targets reduction of stress, but also attempts to resolve the cause of an internal conflict, similar to an emotional decoupling used in trauma therapy. There are already studies on the efficacy of Introvision in chronic neck tension and tinnitus. Please find attached the complete application documents. I would be very happy about a positive vote.

Kind regards

Dr. med. Monika Empl Neurology Consultant